CLINICAL TRIAL: NCT02052713
Title: A Single-Dose, Randomised, Open-Label, Two-Period Crossover Study to Determine the Bioequivalence of the Second Generation Dutasteride and Tamsulosin HCl Combination Capsule in the Fasted State in Healthy Adult Male Subjects
Brief Title: Bioequivalence Study of the Second Generation Dutasteride and Tamsulosin Hydrochloride (HCL) Combination Capsule in Fasted State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 116897
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Urologic Diseases
Keywords: dutasteride; tamsulosin; healthy subject; dutasteride and tamsulosin combination; combination capsule of dutasteride 0.5 mg and tamsulosin HCL 0.4 mg
MeSH Terms: conditions — Urologic Diseases | interventions — Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence AB (Experimental): Subjects will receive Treatment A (commercially available combination of dutasteride 0.5 mg and tamsulosin HCL 0.4 mg) in period 1 and Treatment B (combination of second generation dutasteride 0.5 mg and tamsulosin HCl 0.4 mg combination) in period 2 orally once daily under fasted condition.
  Interventions: Drug: Commercially available combination of dutasteride 0.5 mg and tamsulosin HCL 0.4 mg; Drug: Second generation dutasteride 0.5 mg and tamsulosin HCL 0.4 mg combination capsule
- Sequence BA (Experimental): Subjects will be randomized to receive Treatment B (combination of second generation dutasteride 0.5 mg and tamsulosin HCl 0.4 mg combination) in period 1 and Treatment A (commercially available combination of dutasteride 0.5 mg and tamsulosin HCL 0.4 mg) in period 2 orally once daily under fasted condition.[dutasteride 0.5 mg and tamsulosin HCl 0.4 mg) in period 2 orally once daily under fasted condition.
  Interventions: Drug: Commercially available combination of dutasteride 0.5 mg and tamsulosin HCL 0.4 mg; Drug: Second generation dutasteride 0.5 mg and tamsulosin HCL 0.4 mg combination capsule

INTERVENTIONS:
Drug: Commercially available combination of dutasteride 0.5 mg and tamsulosin HCL 0.4 mg — Commercially available, orange and brown, hard shell capsule, administered orally as a single dose on Day 1 under fasted condition.
Drug: Second generation dutasteride 0.5 mg and tamsulosin HCL 0.4 mg combination capsule — Orange and brown, hard shell capsule, administered orally, as a single-dose on Day 1 under fasted condition.

SUMMARY:
The purpose of this study is to assess the bioequivalence of the second generation dutasteride and tamsulosin hydrochloride (HCL) combination capsule versus currently available commercial combination of dutasteride 0.5 milligram (mg) and tamsulosin HCL 0.4 mg capsule in healthy adult male subjects. Subjects in this study will receive either a single oral dose of the second generation dutasteride 0.5 mg and tamsulosin 0.4 mg combination capsule or a single dose of commercially available combination of dutasteride 0.5 mg and tamsulosin HCL 0.4 mg followed by a 28-day washout period both in fasted state. The study will enroll approximately 92 healthy adult male subjects in order to complete approximately 76 evaluable subjects. The total duration of a subject's involvement in this study is anticipated to be approximately 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males who are 18 to 50 years of age, inclusive.
* Weight range 55 to 95 kg (inclusive) and body mass index (BMI) 18 to 30 kilogram/meter^2 (kg/m^2) (inclusive).
* Healthy subjects defined as individuals who are free from clinically significant illness or disease as determined by the investigator based on their medical history, physical examination, vital signs, laboratory studies, and electrocardiograms (ECGs).
* Single QT interval corrected (QTc) <450 millisecond (msec) or QTc <480 msec in subjects with Bundle Branch Block, no clinically relevant abnormal finding on the screening ECG.
* Serum creatinine <1.5 x upper limit of normal (ULN) at screening.
* Cytochrome P450 enzyme 2D6 (CYP2D6) Extensive Metabolizers only at screening
* Willing and able to give written informed consent.
* Able to swallow and retain oral medication.
* Male subjects with female partners of child-bearing potential must agree to use 1 of the contraception methods. - Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatise (ALP), and bilirubin <=1.5 x ULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

* History of postural hypotension, dizziness, poor hydration, vertigo, vaso-vagal reactions or any other signs and symptoms of orthostasis, which in the opinion of the investigator could be exacerbated by tamsulosin and result in putting the subject at risk of injury.
* History of any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions that could interfere with a subject's safety, or interfere with the subject's ability to follow indications or study procedures, or the interpretation of study results or obtaining informed consent or compliance to study procedures in the opinion of the Investigator or GlaxoSmithKline (GSK) Medical Monitor.
* History of myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, or cerebrovascular accident prior to Screening visit; or diabetes or peptic ulcer disease which is uncontrolled by medical management.
* History of breast cancer or clinical breast examination finding suggestive of malignancy, malignancy within the past 5 years, except for basal cell carcinoma of the skin. Subjects with a prior malignancy who have had no evidence of disease for at least the past 5 years are eligible.
* Prior medical history or evidence of prostate cancer. Subjects with suspicious ultrasound or Digital Rectal Examination (DRE) who have had a negative biopsy within the preceding 6 months and stable prostate specific antigen (PSA) are eligible for the study.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Positive human immunodeficiency virus (HIV) test at screening.
* Use of prescription or non-prescription drugs.
* Strong Cytochrome P450 enzyme 3A4 (CYP3A4) inhibitors (e.g. ketoconazole) and/or strong CYP2D6 inhibitors (e.g. paroxetine) usage throughout the study.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of regular alcohol consumption exceeding 21 drinks/week for men (1 unit is equivalent to 8 gram of alcohol: a half-pint (equivalent to 240 millilitre [mL]) of beer, 1 glass (equivalent to 125 mL) of wine or 1 (equivalent to 25 mL) measure of spirits) within 6 months of screening. Subjects must be able and willing to abstain from beverages and foods containing alcohol 24 hours prior to the first dose of study medication and until the completion of the final PK sample during each period.
* A positive urine drug or alcohol screen result at screening and at Day -1. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids, and benzodiazepines.
* Subjects must be able and willing to stop using of any tobacco or nicotine containing products 24 hours prior to each dose and for the duration of confinement. At the discretion of the Investigator, light smokers (smoking <=10 cigarettes a day) would be considered for the study inclusion.
* The subject has received an investigational product or participated in any other research trial within 6 months or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication or anytime during the study period, exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Previous donation of blood or blood products in excess of 500 mL within a 90 day prior to the first dose of investigational products and the subject agrees not to donate blood during this study.
* History or presence of allergy, intolerance, contraindication or sensitivity to alpha blockers (e.g., tamsulosin), or 5 alpha reductase inhibitors (e.g., dutasteride) or drugs of these therapeutic classes, soya or peanuts, or any ingredients of Combodart, or a history of drug or other allergy (including true sulfonamide allergy) that, in the opinion of the investigator, contraindicates your participation in the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2014-02-19 (Actual); Primary Completion 2014-12-29 (Actual); Study Completion 2014-12-29 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) profile of second generation dutasteride when co-administered with tamsulosin HCL relative to the commercial combination of dutasteride 0.5 mg and tamsulosin HCL 0.4 mg in the fed state to investigate bioequivalence | PK blood samples will be collected at pre-dose, 0, 0.25, 0.50, 0.75, 1, 2, 3, 4, 5, 6, 6.5, 7, 7.5, 8, 10, 12, 16, 24, 48, 72 hour post dose in each period.
  PK parameters include: area under the concentration-time curve from time zero to last time of quantifiable concentration within a subject (AUC [0-t]), and maximum observed concentration (Cmax) as data permit
Composite of PK parameters for tamsulosin HCl when it is co-administered with second generation dutasteride relative to the currently available commercial dutasteride 0.5 mg + tamsulosin HCL 0.4 mg in the fed state to investigate bioequivalence | PK blood samples will be collected at pre-dose, 0, 0.25, 0.50, 0.75, 1, 2, 3, 4, 5, 6, 6.5, 7, 7.5, 8, 10, 12, 16, 24, 48, 72 hour post dose in each period.
  PK parameters include: AUC[0-t]), area under the concentration-time curve from time zero extrapolated to infinite time (AUC[0-infinity]) [defaulting to AUC(0-t)

SECONDARY OUTCOMES:
PK profile of dutasteride | PK blood samples will be collected at pre-dose, 0, 0.25, 0.50, 0.75, 1, 2, 3, 4, 5, 6, 6.5, 7, 7.5, 8, 10, 12, 16, 24, 48, 72 hour post dose in each period.
  PK parameters include: time of occurrence of Cmax (tmax), and negative slope of the terminal phase (lambda) as data permit.
PK profile of tamsulosin HCl | PK blood samples will be collected at pre-dose, 0, 0.25, 0.50, 0.75, 1, 2, 3, 4, 5, 6, 6.5, 7, 7.5, 8, 10, 12, 16, 24, 48, 72 hour post dose in each period.
  PK parameters include: tmax, lambda, and half life (t1/2)
Clinically significant changes in Vital signs measurements to assess safety and tolerability | Baseline (screening) and up to 33 days.
  Vital signs will include blood pressure and pulse rate measurements
Incidence of adverse events (AEs) | Up to 48 days
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Clinical laboratory parameter assessment as a measure of safety and tolerability | Up to 33 days
  Laboratory parameters include: hematology, clinical chemistry and urinalysis.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: Results for study 116897 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116897?search=study&search_terms=116897#rs